CLINICAL TRIAL: NCT05485025
Title: Long Term Prospective Study of Tai Chi Intervention to Delay the Progression of Subjective Cognitive Impairment
Acronym: TIPS
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ruijin Hospital (Other)
Collaborators: Zhangjiagang Aoyang Hospital of Jiangsu Province (Unknown)
Responsible Party: Principal Investigator, Shengdi Chen, Professor, Ruijin Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: TIPS Study
Record Dates: First submitted 2022-07-28; First posted 2022-08-02 (Actual); Last update posted 2022-08-02 (Actual); Status verified 2022-07

CONDITIONS: Subjective Cognitive Impairment
Keywords: subjective cognitive impairment; Tai Chi

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Tai chi training plus group activity (Experimental): Tai chi training: a teacher will give two 60-min lessons per week. Participants will play Tai Chi in the lessons, following teacher's instruction.
  Group activity: a organizer will lead the subjects to participate in group activities, once per quarter.
  Interventions: Behavioral: Tai chi training; Behavioral: Group activity
- Only group activity (Experimental): Group activity: a organizer will lead the subjects to participate in group activities, once per quarter.
  Interventions: Behavioral: Group activity

INTERVENTIONS:
Behavioral: Tai chi training — Tai chi, also called tai chi chuan, is an ancient Chinese form of exercise originally created as a fighting art. It is a kind of gentle physical exercise and stretching, which involves a series of movements performed in a slow, focused manner and accompanied by deep breathing.
  Arms: Tai chi training plus group activity
Behavioral: Group activity — A organizer will lead the subjects to participate in group activities once a quarter. In group activities, there will be popular science lectures and interactive games.

SUMMARY:
This study evaluates the effects of 3 years-Tai Chi exercise intervention on cognitive function in subjects with subjective cognitive impairment (SCI). Participants will be randomized into the Tai chi training group and the control group.

DETAILED DESCRIPTION:
Dementia is a syndrome of impairments of cortical functions caused by brain diseases. More than 55 million people worldwide are currently living with dementia, with nearly 10 million new cases each year. Alzheimer's disease (AD) is the most common form of dementia and may account for 60-70% of patients with dementia. Mild cognitive impairment (MCI) is an intermediate state between normal cognitive aging and dementia. About 10% to 15% of patients with MCI progress to dementia each year. In recent years, studies have found that there is an earlier stage before MCI, that is, the stage of subjective cognitive impairment (SCI). SCI is a stage between normal aging and MCI, which is manifested by the self-reported experience of worsening or more frequent memory loss but not supported by objective evidence. Subjects with SCI are more likely to develop AD. According to the US CDC data, the prevalence of SCI among adults aged 65 years and older is 11.7%. Therefore, it is crucial to find intervention strategies to prevent the progression of SCI to MCI and dementia. However, drug interventions are currently ineffective in the prevention and treatment of such diseases. Based on the synaptic plasticity, more and more studies focus on non-drug interventions. Our research group previously found non-drug interventions (cognitive training, exercise therapy) can effectively delay cognitive decline in the elderly. Therefore, this project plans to conduct a multi-site, randomized, parallel-controlled clinical trial to examine the effect of 3 years-Tai Chi exercise intervention on cognitive function in SCI subjects and to provide a new clinical basis for the prevention and treatment of cognitive disorders.

ELIGIBILITY:
Inclusion Criteria:

1. Male and female participants aged 60 to 75 years (inclusive) at the time of screening;
2. Willing and able to give informed consent by GCP and local guidance;
3. Meets the diagnostic criteria for subjective cognitive impairment (SCI) and the following criteria

   * Subjective decline in memory, rather than other domains of cognition
   * Onset of SCI within the last 5 y
   * Concerns (worries) associated with SCI
   * Feeling of worse performance than others of the same age group
   * Confirmation of cognitive decline by an informant.
4. Have the physical, cognitive, listening, speech, literacy and language skills necessary to participate in all tests;
5. Capable of performing MR.

Exclusion Criteria:

1. Cognitive impairment caused by other reasons (for example) cerebrovascular disease, central nervous system infection, Creutzfeldt-Jakob disease, Huntington's disease, Parkinson's disease, dementia with Lewy bodies, trauma, other physical and chemical factors (drugs, alcohol, CO, etc.), important physical diseases (hepatic encephalopathy, pulmonary encephalopathy, etc.), brain tumor, endocrine diseases (thyroid disease, parathyroid disease), and vitamin deficiency or any other cause of dementia;
2. Abnormal folate, thyroid, and/or vitamin B12 values that cannot be corrected before baseline visit;
3. Major structural brain disease as judged by central MRI Diagnostic Imaging Review Team (eg, ischemic infarcts, subdural hematoma, hemorrhage, hydrocephalus, brain tumors, multiple subcortical ischemic lesions. or a single lesion in a critical region [eg, thalamus]). Mild white matter changes without clinical significance and no more than 2 lacunar infarcts are permitted;
4. Geriatric Depression Scale-15(GDS-15) total score > 7 at screening;
5. MOCA<26 points;
6. CDR global score >0;
7. Hachinski ischemia score >4;
8. During the clinical study, the following drugs are prohibited:

   Acetylcholinesterase inhibitors, N-methyl-D-aspartate (NMDA) antagonists (eg, memantine), central nervous system stimulants, and various medicines that can improve memory or cognition; Antipsychotics
9. Mental illness determined by Diagnostic and Statistical Manual of Mental Disorders (DSM) V criteria, that is unstable within 12 months, or would interfere with study assessments, including schizophrenia or other psychotic disorders, bipolar disorder, severe depression, or delirium.
10. DSM V diagnosis of alcohol or other substance abuse dependence within the last 12 months.
11. History or current diagnosis of significant cardiac arrhythmias, myocardial infarction, transient ischemic attack, or cerebrovascular accident, uncompensated congestive heart failure New York Heart Association class III and IV.
12. Major medical illness or unstable medical condition within 6 months of screening that in the opinion of the investigator may interfere with the participant's ability to comply with study procedures and abide by study restrictions, or with the ability to interpret safety data, including any physical disability (eg. blindness. deafness, non-cognitive related speech impairment, sensory or motor dysfunction) that would prevent completion of study procedures or assessments.
13. Cancer except:

    History of any cancer that has been in remission (no evidence of recurrence) for > 5 years from the screening Participants with basal cell or stage I squamous cell carcinoma of the skin, stable untreated cancer as prostate or meningioma.
14. Active physical activity for 6 months prior to screening.
15. Participants are excluded if they

    1. have participated in any other clinical study within 4 weeks prior to screening visit
    2. have participated in another Tai chi clinical study at any time
    3. plan to take part in another clinical study during this study.
16. The researcher estimates that the subject's compliance is poor, and it is believed that the subject is unlikely to complete the study.

Ages: 60 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 134 (Estimated)
Dates: Start 2022-09 (Estimated); Primary Completion 2026-09 (Estimated); Study Completion 2026-09 (Estimated)

PRIMARY OUTCOMES:
The global cognitive function of SCI subjects. | 36 months
  Repeatable Battery for the Assessment of Neuropsychological Status(RBANS) will be used to assess the global cognitive performance of SCI subjects.

SECONDARY OUTCOMES:
Memory | 18 months and 36 months
  Memory will be assessed using the Auditory verbal learning test-Huashan version (AVLT-H).
Attention | 18 months and 36 months
  Attention will be evaluated by Trial Making Test (TMT).
Executive function | 18 months and 36 months
  Executive function will be evaluated by the Stroop task.
Language | 18 months and 36 months
  Language will be assessed by Boston naming test (30-item version), and Verbal Fluency.
Working memory test | 18 months and 36 months
  Working memory test will be assessed by Number Span Forward and Backward.
Visual spatial ability | 18 months and 36 months
  Visual spatial ability will be assessed by Clock Drawing Test.
Change from baseline in MoCA score | 18 months and 36 months
  Change from baseline in Montreal Cognitive Assessment (MoCA) score.
Change from baseline in CDR score | 18 months and 36 months
  Change from baseline in Clinical Dementia Rating (CDR) Scale score.
Activities of daily living | 18 months and 36 months
  Activities of daily living will be assessed by functional activities questionnaire (FAQ).
Anxiety | 18 months and 36 months
  Anxiety will be assessed by Hamilton Anxiety Rating Scale (HAMA).
Depression | 18 months and 36 months
  Depression will be assessed by Hamilton Depression Rating Scale (HAMD).
Sleep | 18 months and 36 months
  Sleep will be assessed by Pittsburgh Sleep Quality Index (PSQI).
Brain activity | 36 months
  Detecting changes associated with blood flow by fMRI.
Neurodegeneration in brain structures | 36 months
  Brain atrophy will be assessed by Magnetic Resonance Volume Imaging.
Gut microbiota | 18 months and 36 months
  Gut microbiota will be assessed by 16S rRNA sequencing.
Blood biomarkers | 18 months and 36 months
  Inflammatory factors (FGF basic、Eotaxin、G-CSF、GM-CSF、IFN-γ、IL-1β、IL-1ra、IL-2、IL-4、IL-5、IL-6、IL-7、IL-8、IL-9、IL-10、IL-12 (p70)、IL-13、IL-15、IL-17、IP-10、MCP-1 (MCAF)、MIP-1α、MIP-1β、PDGF-BB、RANTES、TNF-α、VEGF) will be measured by Bio-Plex Human Cytokine Assays. Nfl, Aβ40, Aβ42,T-tau, p-tau
Gait and Hand writing Task | 18 months and 36 months
  Using wearable sensors to assess gait and hand writing task.
Incidence of SCI converted to MCI and Alzheimer's disease. | 36 months
  The 3-year incidence of MCI and AD in each group will be compared.

CONTACTS AND LOCATIONS:
Locations (1):
- Shanghai Jiao Tong University School of Medicine Affiliated Ruijin Hospital, Shanghai, China

IPD SHARING:
Plan to Share IPD: No